CLINICAL TRIAL: NCT02025231
Title: Image Guided Reirradiation of High-grade Glioma - a Phase I/II Dose Escalation Study
Brief Title: Image Guided Reirradiation of High-grade Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Principal Investigator, Søren Møller, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RH ReRT 2011; H-2-2011-092 (Registry Identifier: Capital Region Commitee on Health Research Ethics)
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Malignant Glioma; Glioblastoma
Keywords: reirradiation; recurrent glioma; positron emission tomography; amino acid tracer
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External beam radiotherapy (Experimental): Hypofractionated external beam radiation delivered in 4 different sequential dose/fractionation groups.
  Interventions: Radiation: External beam radiotherapy

INTERVENTIONS:
Radiation: External beam radiotherapy — Study group 1: 3.5 Gray x 10, 5 fractions per week. Study group 2: 3.5 Gray x 10 + 7 Gray boost to biological target volume, 5 fractions per week. Study group 3: 5.9 Gray x 10, 5 fractions per week. Study group 4 (planning target volumes: 100 millilitres - 300 millilitres): 3.5 Gray x 10, 5 fractions per week. Phase II dosis: to be chosen based on results of phase I study.

SUMMARY:
The purpose of the study is to evaluate the short- and long term toxicity of radiotherapy to patients with recurrent high-grade glioma who have previously received radiotherapy and to determine the best dose and treatment regimen. Positron emission tomography (PET) using an amino acid tracer, 18-fluoro-ethyltyrosine (18F-FET), is used for target delineation.The study examines, in four sequential treatment groups, the effect of dose, hypofractionation and treatment volume on toxicity. Upon completion of the phase I part, the study progresses to phase II where the best dose- and treatment regimen will be chosen for treatment.

ELIGIBILITY:
Inclusion Criteria:

* recurrent high-grade glioma
* previous focal radiotherapy for high-grade glioma
* no standard treatment options available/indicated
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1 or 2
* life expectancy > 3 months
* hemoglobin value > 6 mmol/l (transfusion permitted)
* able to understand oral and written Danish

Exclusion Criteria:

* disseminated recurrent disease
* infection or wound dehiscence or other pathological condition in meninges/skull/scalp
* symptoms of elevated intracranial pressure
* very early recurrence following primary radiotherapy (< or equal to 3 months)
* contraindications to magnetic resonance imaging (MRI) or positron emission tomography (PET)
* other previous radiotherapy to the brain than primary course of irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | One year
  Early (<4 weeks) and late (> 4 weeks) toxicity evaluated by Common Toxicity Criteria ver. 3.0 at multiple time points up to one year after treatment. (for phase I part of the study)
Diagnostic precision of 18F-FET-PET imaging in recurrent high-grade glioma | Approximately one to two weeks prior to radiotherapy
  Diagnostic accuracy (positive- and negative predictive value) of 18F-FET-PET guided biopsies (optional procedure) in patients who will receive reirradiation for recurrent high-grade glioma in the study. (for phase I part of the study).
Time to neurocognitive decline | Up to one year
  Time to neurocognitive decline assessed using a test battery comprised of validated tests at multiple time points. (for phase II part of the study)
Time to progression | Up to one year
  Time to disease progression evaluated by RANO (Response Assessment in Neuro-Oncology) criteria (for phase II part of the study).

SECONDARY OUTCOMES:
Value of 18F-FET-PET in reirradiation of high-grade glioma | One year
  Prognostic value of 18F-FET-PET scan at baseline, value of 18F-FET-PET as an early response marker and correlations between 18F-FET-PET scans and magnetic resonance imaging.
Objective response rate | Up to one year
  Rate of objective tumor responses following treatment evaluated by RANO criteria and by 18F-FET-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Svend Aage Engelholm, MD, Study Chair — Department of Radiation Oncology, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen Ø
Locations (2):
- Department of Radiation Oncology, Rigshospitalet, Copenhagen, Denmark
- Skånes universitetssjukhus, Lund, Sweden